CLINICAL TRIAL: NCT01409317
Title: Neural Predictors and Longitudinal Neural Correlates of Clinical Improvement After Standard or Deep Transcranial Magnetic Stimulation in Major Depression: A Randomized Study
Brief Title: Neural Predictors and Longitudinal Neural Correlates of Deep Transcranial Magnetic Stimulation for Treating Major Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, MARCELO T. BERLIM, Director, Neuromodulation Research Clinic, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTMS-ERB11/28-2011
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depression; Functional Magnetic Resonance Imaging; Deep Transcranial Magnetic Stimulation; Repetitive Transcranial Magnetic Stimulation; rTMS; DTMS; fMRI; Randomized, Sham-Controlled Trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Transcranial Magnetic Stimulation (Experimental)
  Interventions: Device: Deep Transcranial Magnetic Stimulation
- Repetitive Transcranial Magnetic Stimulation (Active Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation — DTMS will be administered according to the following parameters: 18 Hz in 84 trains of 2 seconds duration, with 20 seconds inter-train interval (3,024 pulses per session) at 120% of the resting motor threshold
  Arms: Deep Transcranial Magnetic Stimulation
Device: Repetitive Transcranial Magnetic Stimulation — rTMS will be administered according to the following parameters: 18 Hz in 84 trains of 2 seconds duration, with 20 seconds inter-train interval (3,024 pulses per session) at 120% of the resting motor threshold.
  Arms: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Standard high frequency repetitive transcranial magnetic stimulation (HF-TMS) is a noninvasive method to activate or de-activate neurons in superficial regions of the brain through the induction of weak electric currents in the brain tissue produced by rapidly changing magnetic fields. Studies have generally shown standard HF-TMS to be effective in treating major depressive disorder (MDD), although treatment effects are often highly variable and there are several negative trials in the specialized literature. One reason for these discrepant results might be that standard HF-TMS only enables direct stimulation of superficial brain areas and, consequently, it is possible that the stimulation of deeper and more widespread brain regions could produce superior and more reliable results. Recently, a novel form of HF-rTMS (called deep transcranial magnetic stimulation or DTMS), that allows direct stimulation of much larger and deeper brain regions, has also been shown to be effective and safe in treating MDD. Neuroimaging studies have shown that standard HF-rTMS directly affects several superficial areas of the brain, but to date there is no data on the brain effects of DTMS. Thus, this study aims to explore, for the first time, the brain effects of DTMS in MDD. More specifically, we, the investigators, hope to identify possible neural predictors of clinical improvement after DTMS and also clarify the impact of DTMS in the brain activity over time. In this study, DTMS will be applied over the left side of the front of the head (a region known as the 'prefrontal cortex'), and will be compared with standard HF-TMS in terms of its effectiveness and brain effects. For this, subjects with at least moderate MDD will be randomized to receive daily DTMS or standard HF-rTMS treatment for 4 weeks, and will undergo functional magnetic resonance imaging (fMRI) before and after treatment. fMRI is a neuroimaging technique that allows us to measure which areas of the brain are more or less 'active' in response to specific stimuli at a particular time. During the fMRI sessions, we will use a validated cognitive task on working memory. Our results could eventually lead us, among other things, to identify which depressed patients would be best candidates for receiving either standard HF-rTMS or DTMS, and which areas of the brain should be targeted by these neuromodulation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a current major depressive disorder (according to the Diagnostic and Statistical Manual, Fourth Edition, Text Revision [DSM-IV-TR]) that has not improved after ≥ 1 but ≤ 3 adequate antidepressant trial(s) in the current episode
* Baseline score ≥ 21 on the HAM-D21
* Stable medication regimen (> 4 weeks)

Exclusion Criteria:

* Psychotic features in the current episode
* Lifetime history of psychotic disorders and/or bipolar I or II disorders
* Substance or alcohol abuse/dependence in the past 6 months
* Lifetime history of a major neurological disease (e.g., Parkinson's, stroke)
* Uncontrolled medical disease (e.g., cardiovascular, renal)
* Pregnancy and/or lactation
* Presence of a specific contraindication for DTMS/rTMS/MRI (e.g., personal history of epilepsy, metallic head implant, cardiac pacemaker)
* Personal history of abnormal brain MRI findings

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
21-item Hamilton Depression Rating Scale (HAM-D21) | week 5
  Pre-post neuromodulation changes on HAM-D21 scores

SECONDARY OUTCOMES:
21-item Hamilton Depression Rating Scale (HAM-D21) | week 5
  Response to treatment is defined as a ≥ 50% reduction in the scores of the HAM-D21. Remission is defined as a HAM-D21 score ≤ 8.
Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) | week 5
  Response is defined as a ≥ 50% reduction in the scores of the QIDS-SR. Remission is defined as a QIDS-SR score ≤ 5.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo T. Berlim, MD, MSc, Principal Investigator — McGill University & Douglas Mental Health University Institute
Locations (1):
- Neuromodulation Research Clinic, Douglas Mental Health University Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Levkovitz Y, Roth Y, Harel EV, Braw Y, Sheer A, Zangen A. A randomized controlled feasibility and safety study of deep transcranial magnetic stimulation. Clin Neurophysiol. 2007 Dec;118(12):2730-44. doi: 10.1016/j.clinph.2007.09.061. Epub 2007 Oct 30. PMID 17977787
- [Background] Levkovitz Y, Harel EV, Roth Y, Braw Y, Most D, Katz LN, Sheer A, Gersner R, Zangen A. Deep transcranial magnetic stimulation over the prefrontal cortex: evaluation of antidepressant and cognitive effects in depressive patients. Brain Stimul. 2009 Oct;2(4):188-200. doi: 10.1016/j.brs.2009.08.002. Epub 2009 Sep 16. PMID 20633419
- [Background] Isserles M, Rosenberg O, Dannon P, Levkovitz Y, Kotler M, Deutsch F, Lerer B, Zangen A. Cognitive-emotional reactivation during deep transcranial magnetic stimulation over the prefrontal cortex of depressive patients affects antidepressant outcome. J Affect Disord. 2011 Feb;128(3):235-42. doi: 10.1016/j.jad.2010.06.038. Epub 2010 Jul 21. PMID 20663568